CLINICAL TRIAL: NCT00888277
Title: Neuropsychological Assessments in the Multiple Sclerosis Clinic
Brief Title: Bayer/Cognitive Assessments With Multiple Sclerosis Subjects
Status: Completed | Type: Observational
Sponsor: University of Louisville (Other)
Collaborators: Bayer Healthcare Pharmaceuticals, Inc./Bayer Schering Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: UofL IRB # 09.0167; OICN 090742
Record Dates: First submitted 2009-04-22; First posted 2009-04-27 (Estimated); Last update posted 2013-11-04 (Estimated); Status verified 2013-10

CONDITIONS: Multiple Sclerosis, Relapsing-remitting; Multiple Sclerosis, Secondary Progressive
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is designed to identify a brief screening evaluation for MS patients that is sensitive and specific to the MS population and which correlates with the findings of our standard-of-care neuropsychological assessments.

DETAILED DESCRIPTION:
Seventy five randomly identified patients will be evaluated. Consenting patients will perform a Symbol Digit Modalities Test (SDMT) and have the MS Center´s standard neuropsychological assessment performed. Tests comprising the standard assessment will be the RBANS (Randolph, 1998), Multiscore Depression Inventory, Cross and Clock Drawings. The selfreported Beck Depression Inventory (BDI-II) will also be obtained. An Expanded Disability Status Scale (EDSS) will be recorded for each patient. The RBANS consists of six scales labeled (1) Immediate Memory, (2) Visuospatial/ Constructional, (3) Language, (4) Attention, (5) Delayed Memory, and (6) Total. Depression will be assessed by the BDI and the MultiScore Depression Inventory.

The SDMT will be administered using standard instructions either orally or in writing. Use of the established norms for the SDMT will be used to determine if the MS patient is demonstrating some cognitive dysfunction. Scores less than 1.0 to 1.5 standard deviations below mean are suggestive of cerebral dysfunction. The results will be controlled for age, gender, and educational level.

Additionally, the results of the 75 patient assessments will be reviewed to see the concordance between the results of the SDMT and the Neuropsychological Battery. The association of cognitive dysfunction as identified by the SDMT will be correlated with each of the six RBANS scales and other parameters of the cognitive aspects of the Battery. Statistical analysis will determine the sensitivity and specificity of the SDMT in determining abnormalities as well as an optimum cutpoint. This analysis will indicate possible cognitive problems and the need for further testing and, potentially, intervention.

ELIGIBILITY:
Inclusion Criteria:

* EDSS at last visit ≤ 7.0
* Relapsing/Remitting or Secondary Progressive MS

Exclusion Criteria:

* Severe Depressive Illness: Beck Depression Inventory Score > 55.
* Unable to read with/without glasses- Visual Acuity better than or equal to 20/60 in one eye.
* Unwilling to sign Informed Consent.
* Evidence on clinical examination of severe dementia at discretion of evaluating neurologist.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subjects will be recruited from patients diagnosed with MS at the University of Louisville Neurologists PCS.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2009-05; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
SDMT correlation with the findings on the Neuropsychological Battery. The Neuropsychological Battery will confirm that the SDMT is sensitive and specific in identifying MS patients with cognitive findings. | 1 year

SECONDARY OUTCOMES:
SDMT association with the BDI. The SDMT will be independent of depression. | 1 year
Overlap of Depression with Cognitive Dysfunction. There will still be identified a high percentage of patients having both cognitive and depressive symptoms. | 1 year
Lack of association of Cognitive Dysfunction with the Physical Scales of the EDSS. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Richard Kirzinger, MD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, Louisville, Kentucky, United States